CLINICAL TRIAL: NCT05915195
Title: Effects of Postural and Kinesthetic Awareness on Static Standing Balance and Planter Pressure by Using PoData Stabiliometric Plate in Stroke
Brief Title: Effects of Postural and Kinesthetic Awareness on Static Standing Balance in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Safa Saleem, Prinicipal Investigator, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-70-02-2023
Record Dates: First submitted 2023-04-14; First posted 2023-06-22 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Chronic Stroke
Keywords: stroke; static balance; plantar pressure; postural and kinestetic awareness; PoData Stabiliometeric plate
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Physical Therapy (Active Comparator): routine physical therapy including range of motion exercises (Active assisted), stretching exercises, strengthening and positioning. Daily session was of 1 hour, 5 times weekly for 6 weeks.
  Interventions: Other: Routine Physical Therapy
- Routine Physical Therapy and Postural and Kinesthetic Awareness (Experimental): routine physical therapy and additionally postural and kinesthetic Awareness in front of mirror by emphasizing proper body positioning, movements & balance in sitting and standing position by using interoceptive and exteroceptive reinforcement (verbal, tactile & visual).
  Interventions: Other: Postural and Kinesthetic Awarness

INTERVENTIONS:
Other: Postural and Kinesthetic Awarness — Firstly, patient performed therapeutic activities/exercise to achieve balance in sitting position using chair with arm rest and with planted feet then progressed to sitting on chair without arm rest with proper feet placement. Once the patient achieved balance in sitting on chair then shifted to sitting on the stool and later standing in parallel bar that leads to balance training in independent standing.
  Other Names: Experimental Group
  Arms: Routine Physical Therapy and Postural and Kinesthetic Awareness
Other: Routine Physical Therapy — Range of motion exercises (Active assisted), stretching exercises, strengthening and positioning.
  Other Names: Control Group
  Arms: Routine Physical Therapy

SUMMARY:
The goal of this randomized controlled trial is to check the effects of postural and kinesthetic awareness on static standing balance in chronic stoke patients. Participants will be divided into two equal groups. One group will receive routine physical therapy while other group will receive postural and kinesthetic awareness in addition to routine physical therapy.

DETAILED DESCRIPTION:
To determine effects of Postural and kinesthetic awareness on plantar pressure and static standing balance in chronic stroke patients. The study was conducted at the University of Lahore Teaching Hospital in the Department of Pediatric Physical Therapy & Neuro Rehabilitation Center. Total 62 stroke patients with visual spatial neglect were enrolled in this study, patients were equally assigned into control and experimental group. Control group received routine physical therapy while experimental group received routine physical therapy and postural and kinesthetic awareness program. Static component of berg balance scale and PoData Stabiliometeric plate was used for measurement of balance and plantar pressure respectively

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke patient
* Both genders
* Age: 45-60 years
* 9 score or higher on static part of Berg Balance Scale
* Level 1 and 2 of Modified Ashworth Scale
* 24 or more score on Mini mental state scale

Exclusion Criteria:

* Patients with

  * Psychological diseases
  * Dementia
  * Orthopedic disorders
  * Any insufficiency that can influence balance

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Static Component of Berg Balance Scale | 6 months
  Static component of Berg Balance Scale was used to measure static standing balance. Total score of berg balance scale is 56. A score of 56 indicates functional balance.A score of < 45 indicates individuals may be at greater risk of falling.
PoData Stabiliometric Plate | 6 months
  PoData stabiliometric plate was used for the static plantar pressure evaluation. It recorded statistics of plantar pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Sameed Liaquat, MSPTN, Principal Investigator — University of Lahore
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rauf W, Sarmad S, Liaqat S, Saleem S, Jawad M, Ahad M. Effects of postural and kinesthetic awareness on static standing balance and plantar pressure in chronic stroke: a randomized controlled trial. J Pak Med Assoc. 2024 Oct;74(10):1755-1760. doi: 10.47391/JPMA.10538. PMID 39407366